CLINICAL TRIAL: NCT05668858
Title: A Phase Ib/II Clinical Study of SI-B001+SI-B003 Dual-drug No-combination or Combined Chemotherapy in Patients With Locally Advanced or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of SI-B001+SI-B003± Chemotherapy in Patients With Locally Advanced or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001-SI-B003-201
Record Dates: First submitted 2022-12-09; First posted 2022-12-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants will receive treatment during the first cycle. Participants with clinical benefits received more cycles of additional therapy. Administration will be discontinued due to disease progression or occurrence of intolerable toxicity or other reasons.
  Interventions: Drug: SI-B001; Drug: SI-B003

INTERVENTIONS:
Drug: SI-B001 — Administration by intravenous infusion
Drug: SI-B003 — Administration by intravenous infusion

SUMMARY:
Phase Ib: To observe the safety and tolerability of SI-B001+SI-B003 in combination and to identify RP2D in locally advanced or metastatic head and neck squamous cell carcinoma indications. Initial efficacy, pharmacokinetic characteristics and immunogenicity were evaluated. Phase II: To evaluate the efficacy of SI-B001+SI-B003 two-drug combination chemotherapy. Safety and tolerance, PK/PD, immunogenicity were evaluated.

DETAILED DESCRIPTION:
Phase Ib: To observe the safety and tolerability of SI-B001+SI-B003 combination and to determine the recommended dose (RP2D) for Phase II clinical studies in locally advanced or metastatic head and neck squamous cell carcinoma indications. To evaluate the initial efficacy, pharmacokinetic characteristics and immunogenicity of SI-B001+SI-B003 in patients with locally advanced or metastatic head and neck squamous cell carcinoma. Phase II: To evaluate the efficacy of SI-B001+SI-B003 dual-agent chemotherapy in patients with locally advanced or metastatic head and neck squamous cell carcinoma. The safety, tolerability, PK/PD and immunogenicity of SI-B001+SI-B003 combined chemotherapy in patients with locally advanced or metastatic head and neck squamous cell carcinoma were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Histologically or cytologically confirmed head and neck squamous cell carcinoma occurring only in the oral cavity, oropharynx, hypopharynx, and larynx;
6. Agree to provide archived tumor tissue specimens or fresh tissue samples from primary or metastatic lesions;
7. Must have at least one measurable lesion as defined by RECIST v1.1;
8. Performance status score: ECOG ≤1;
9. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50%;
11. Organ function levels must meet the requirements;
12. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
13. Urine protein ≤1+ or ≤1000 mg/24h;
14. Female subjects of childbearing potential or male subjects with partners of childbearing potential must use highly effective contraception from 7 days before the first dose until 24 weeks after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Squamous cell carcinoma originating from the nasopharynx, salivary glands, nasal sinuses, skin, or with an unknown primary site;
2. For Phase II patients, either: a) those suitable for and willing to undergo local therapy; or b) those who have received systemic chemotherapy, excluding chemotherapy administered as part of multimodal treatment for locally advanced disease;
3. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (leptomeningeal metastases) and/or spinal cord compression;
4. Participation in any other clinical trial within 4 weeks prior to the administration of this trial's investigational product (based on the last dose date);
5. Receipt of chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, or other antitumor treatments within 4 weeks before the first dose of the study drug;
6. Major surgery (as defined by the investigator) within 4 weeks prior to the first dose;
7. Requirement for systemic corticosteroids or immunosuppressive therapy within 2 weeks before the study drug administration;
8. Pulmonary diseases graded as ≥Grade 3 according to NCI-CTCAE v5.0; current or history of interstitial lung disease (ILD);
9. Active infection requiring intravenous anti-infective therapy;
10. Prior immunotherapy leading to ≥Grade 3 immune-related adverse events (irAE) or ≥Grade 2 immune-related myocarditis;
11. Use of live attenuated vaccines within 4 weeks before the first dose of the study drug;
12. Use of immunomodulatory drugs (including but not limited to thymosin, interleukin-2, interferon, etc.) within 14 days before the first dose of the study drug;
13. Patients at risk of active autoimmune diseases or with a history of autoimmune diseases;
14. History of other malignancies within 5 years before the first dose;
15. Positive for human immunodeficiency virus (HIV) antibodies, active tuberculosis, active hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection;
16. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg);
17. History of severe cardiovascular or cerebrovascular diseases;
18. Previous allogeneic stem cell, bone marrow, or organ transplantation;
19. Patients with significant serous cavity effusion, symptomatic effusion, or poorly controlled effusion;
20. History of hypersensitivity to recombinant humanized antibodies or any excipients of SI-B001 or SI-B003;
21. History of severe infusion reactions (CTCAE Grade ≥3) to antibody therapy;
22. History of autologous or allogeneic stem cell transplantation;
23. Pregnant or lactating women;
24. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B001+SI-B003.
Phase Ib: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Dose Limited Toxicity (DLT) | Up to approximately 24 months
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).
Phase Ib: Maximum Tolerated dose (MTD) or maximum administered dose (MAD) | Up to approximately 24 months
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Phase II: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase Ib/II: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of SI-B001+SI-B003. The type, frequency and severity of TEAE will be evaluated during the treatment of SI-B001+SI-B003.
Phase Ib/II: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib/II: Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib/II: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of SI-B001+SI-B003 to the first date of either disease progression or death, whichever occurs first.
Phase Ib/II: Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of SI-B001+SI-B003 will be investigated.
Phase Ib/II: Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of SI-B001+SI-B003 will be investigated.
Phase Ib/II: T1/2 | Up to approximately 24 months
  Half-life (T1/2) of SI-B001+SI-B003 will be investigated.
Phase Ib/II: AUC0-t | Up to approximately 24 months
  Blood concentration - Area under time line.
Phase Ib/II: CL | Up to approximately 24 months
  To study the serum clearance rate of SI-B001+SI-B003 per unit time.
Phase Ib/II: Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of SI-B001+SI-B003 prior to the next dose will be administered.
Phase Ib/II: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-SI-B001, SI-B003 antibody (ADA) will be evaluated.
Phase Ib/II: Neutralizing antibody (Nab) | Up to approximately 24 months
  Incidence and titer of Nab of SI-B001 and SI-B003 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, PHD, Principal Investigator — Shanghai Oriental Hospital
Locations (1):
- Shanghai Oriental Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No